CLINICAL TRIAL: NCT01226498
Title: Effects of Duration of Stored Red Blood Cell Transfusion on Physiological Parameters and Inflammatory Mediators in Healthy Adult Volunteers
Brief Title: Effects of Blood Transfusion in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Warren M. Zapol, MD, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2010P000961
Record Dates: First submitted 2010-10-14; First posted 2010-10-22 (Estimated); Last update posted 2014-01-30 (Estimated); Status verified 2014-01

CONDITIONS: Blood Transfusion, Autologous
Keywords: Blood Transfusion, Autologous; Blood Preservation/adverse effects; Blood Transfusion/adverse effects; Endothelium, Vascular/physiopathology; Inflammation Mediators

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fresh blood auto-transfusion (Experimental)
  Interventions: Procedure: Red blood Cells auto-transfusion
- Old blood auto-transfusion (Experimental)
  Interventions: Procedure: Red blood Cells auto-transfusion

INTERVENTIONS:
Procedure: Red blood Cells auto-transfusion — Withdrawal from 10 Healthy volunteers of one unit of red blood cells and auto-transfusion after 3 days for one arm of the study, after 40 days for the other. Participants are enrolled in both arms of the study.

SUMMARY:
The objective of this study is to assess effects of the storage of PRBC on endothelial function, inflammation and platelet activation in healthy volunteers

DETAILED DESCRIPTION:
The objective of this study is to assess effects of the storage of PRBC on endothelial function, inflammation and platelet activation in healthy volunteers.

The present study consists of two parts. During one phase of the study, 10 healthy human volunteers will donate a unit of blood, which will be leukoreduced and stored in Additive Solutions-1 (AS-1), and then transfused back to the subjects after 2 days of storage at 4º C in the MGH Blood Bank. The other part of the study consists in the collection of a unit of blood from the same volunteers, but which will be transfused back to the same subject after 40 days of storage. There will be a break of 2 week period in between these 2 study phases. The order of these 2 study parts will be randomized.

We hypothesize that old red blood cells stored under conventional conditions may trigger a complex, pro-inflammatory, pro-thrombotic and vasoconstriction response. We will compare the response to PRBC stored for 2 days with the response to PRBC stored for 40 days in the same healthy volunteers. We will monitor/measure the following markers/parameters:

1. Endothelium-mediated changes in vascular (arterial) tone
2. Tissue oxygen saturation will be continuously assessed during and after blood transfusion
3. Hemolysis as quantified by changes in plasma haptoglobin level, plasma free hemoglobin, LDH level, bilirubin level, iron level, ferritin, and transferrin
4. Changes of plasma and red blood cell levels of circulating nitrate, nitrite, RXNO, RNNO, NO-heme
5. Concentration of cytokines, such as IL-6, IL-8, IL-10, IL-12, TNF, IFN-γ
6. Activation of platelets through circulating P-selectin expression on platelets
7. Activation of inflammatory lipid mediators
8. Changes in gene expression profiling analyzing RNA microarray of circulating leukocytes

ELIGIBILITY:
Inclusion Criteria:

* Have a photo ID
* Body mass index (BMI) <25 kg/m2 and >18 kg/m2
* Fasting for 8 hours prior to enrollment in the study (a sip of water or brushing teeth in the morning are allowed)
* Feel well the day of blood donation
* Normal physical exam and normal blood test as indicated:
* WBC 4.5-11.0 th/cmm
* HGB 12.5-17.5 gm/dl
* PLT 150-400 th/cumm
* Plasma Sodium 135-145 mmol/L
* Plasma Potassium 3.4-4.8 mmol/L
* Plasma Chloride 98-108 mmol/L
* Plasma Carbon Dioxide 23.0-31.9 mmol/L
* Plasma Urea Nitrogen 8-25 mg/dl
* Plasma Creatinine 0.60-1.50 mg/dl
* Plasma Glucose 70-110 mg/dl
* Transaminase-SGPT 10-55 U/L
* Transaminase-SGOT 10-40 U/L

Exclusion Criteria:

* Psychiatric disturbances such as anxiety, depression, schizophrenia requiring pharmacological treatment or hospitalization in the last year
* Systemic disease with or without any functional limitation
* controlled hypertension
* controlled diabetes without systemic effects
* Pregnancy determined by urine pregnancy test, detecting presence of human chorionic gonadotropin (hCG), or less than six weeks postpartum
* Active smoking. Volunteers may be enrolled if they quit smoking for more than 1 year
* Excess alcohol use: more than ½ L/day of wine consumption or equivalent
* Any current use of a medication other than: Over-the-counter oral medications, herbal remedies, nutritional supplements, and oral contraceptives
* Antibiotic use within 48 hours of blood donation
* Use of NSAIDS, corticosteroids, aspirin during the past 7 days
* Dental work within 24 hours prior to the donation
* Received or donated blood in the last 4 months
* Have had any forms of cancer with the exceptions of basal cell skin cancer or treatment for in situ cervical cancer
* Currently enrolled in another research study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2010-07; Primary Completion 2010-11 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Endothelial function | Baseline
Endothelial function | 10 min after transfusion
Endothelial function | 1h after transfusion
Endothelial function | 4h after transfusion

SECONDARY OUTCOMES:
Hemolysis | Baseline
NO metabolites | Baseline
Concentration of cytokines | Baseline
Activation of platelets | Baseline
Activation of inflammatory lipid mediators | Baseline
Changes in gene expression | Baseline
Hemolysis | 10 min after transfusion
NO metabolites | 10 min after transfusion
Concentration of cytokines | 10 min after transfusion
Activation of platelets | 10 min after transfusion
Activation of inflammatory lipid mediators | 10 min after transfusion
Changes in gene expression | 10 min after transfusion
Hemolysis | 1h after transfusion
NO metabolites | 1h after transfusion
Concentration of cytokines | 1h after transfusion
Activation of platelets | 1h after transfusion
Activation of inflammatory lipid mediators | 1h after transfusion
Changes in gene expression | 1h after transfusion
Hemolysis | 2h after transfusion
NO metabolites | 2h after transfusion
Concentration of cytokines | 2h after transfusion
Activation of platelets | 2h after transfusion
Activation of inflammatory lipid mediators | 2h after transfusion
Changes in gene expression | 2h after transfusion
Hemolysis | 4h after transfusion
NO metabolites | 4h after transfusion
Concentration of cytokines | 4h after transfusion
Activation of platelets | 4h after transfusion
Activation of inflammatory lipid mediators | 4h after transfusion
Changes in gene expression | 4h after transfusion

CONTACTS AND LOCATIONS:
Overall Officials: Warren M Zapol, MD, Principal Investigator — Massachusetts General Hospital, DACCPM
Locations (1):
- Massachusetts General Hospital (MGH), Boston, Massachusetts, United States

REFERENCES:
- [Background] Hendrickson JE, Hillyer CD. Noninfectious serious hazards of transfusion. Anesth Analg. 2009 Mar;108(3):759-69. doi: 10.1213/ane.0b013e3181930a6e. PMID 19224780
- [Background] Koch CG, Li L, Sessler DI, Figueroa P, Hoeltge GA, Mihaljevic T, Blackstone EH. Duration of red-cell storage and complications after cardiac surgery. N Engl J Med. 2008 Mar 20;358(12):1229-39. doi: 10.1056/NEJMoa070403. PMID 18354101
- [Background] Bennett-Guerrero E, Veldman TH, Doctor A, Telen MJ, Ortel TL, Reid TS, Mulherin MA, Zhu H, Buck RD, Califf RM, McMahon TJ. Evolution of adverse changes in stored RBCs. Proc Natl Acad Sci U S A. 2007 Oct 23;104(43):17063-8. doi: 10.1073/pnas.0708160104. Epub 2007 Oct 11. PMID 17940021
- [Background] Cardillo C, Kilcoyne CM, Cannon RO 3rd, Panza JA. Interactions between nitric oxide and endothelin in the regulation of vascular tone of human resistance vessels in vivo. Hypertension. 2000 Jun;35(6):1237-41. doi: 10.1161/01.hyp.35.6.1237. PMID 10856270
- [Background] Panza JA, Casino PR, Kilcoyne CM, Quyyumi AA. Role of endothelium-derived nitric oxide in the abnormal endothelium-dependent vascular relaxation of patients with essential hypertension. Circulation. 1993 May;87(5):1468-74. doi: 10.1161/01.cir.87.5.1468. PMID 8491001
- [Background] Gladwin MT, Lancaster JR Jr, Freeman BA, Schechter AN. Nitric oxide's reactions with hemoglobin: a view through the SNO-storm. Nat Med. 2003 May;9(5):496-500. doi: 10.1038/nm0503-496. No abstract available. PMID 12724752
- [Background] Nagasaka Y, Fernandez BO, Garcia-Saura MF, Petersen B, Ichinose F, Bloch KD, Feelisch M, Zapol WM. Brief periods of nitric oxide inhalation protect against myocardial ischemia-reperfusion injury. Anesthesiology. 2008 Oct;109(4):675-82. doi: 10.1097/ALN.0b013e318186316e. PMID 18813047